CLINICAL TRIAL: NCT03048435
Title: Feasibility and Acceptability of Measuring Cervical Cancer Specific Patient-Reported Outcomes in Clinical Practice
Brief Title: Cervical Ca PROs in Clinical Practice
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: OCREB 16-055
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Cervical Cancer; Radiation Therapy
Keywords: Cervical Cancer; Patient Reported Outcomes; Radiation Therapy; EORTC QLQ-CX24; Quality of Life
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cervical Cancer Patients: Adult, English-speaking cervical cancer patients, who have been treated with curative intent chemo-radiotherapy.
  Interventions: Other: EORTC QLQ CX-24
- Oncologist: Oncologists who treat cervix cancer, with at least one consenting patient enrolled in the study.
  Interventions: Other: Physician Feedback Form

INTERVENTIONS:
Other: EORTC QLQ CX-24 — Disease specific Patient Reported Outcome measurement tool developed by the European Organization for Research and Treatment of Cancer (EORTC). This questionnaire covers symptoms common to women with cervical cancer and captures the impact of disease and/or treatment on domains including: urologic and gastro-intestinal symptoms, sexual functioning and body image.
  Other Names: Quality of Life questionnaire
  Groups: Cervical Cancer Patients
Other: Physician Feedback Form — This Feedback form to be completed by oncologists who have had at least one consenting patient participating in this study.
  Groups: Oncologist

SUMMARY:
Concurrent chemo-radiotherapy followed by intracavitary brachytherapy is standard of care for patients with locally advanced cervical cancer. Although curative, this treatment is challenging and leaves a significant proportion of women with severe toxicity, negatively impacting their quality of life. Although most recover over time, a proportion of women do not. Therefore, evaluation of quality of life becomes increasingly more important as cancer specific outcomes improve. One such method is through patient-reported outcomes (PROs), defined as "any report coming directly from the patient about a health condition and its treatment." This prospective multi-institutional study, involving the Princess Margaret (PM), Odette Regional Cancer Centre(ORCC) and Royal Victoria Regional Health Center (RVH), will assess to feasibility and acceptability of integrating a cervical cancer specific PRO measurement tool into clinical practice. Cervical cancer patients coming for follow-up appointments will be asked to complete the EORTC QLQ-CX24, a validated cervical cancer specific PRO questionnaire. At the end of the study period, Feedback Forms will be completed by participating patients and health care providers to obtain their perspectives regarding the feasibility and acceptability of incorporating the instrument into clinical practice. Future directions include designing an electronic platform and expanding its use in cervical cancer clinics provincially and nationally. The data collected should help identify disease-related symptoms, treatment-related toxicities, facilitate patient-physician communication, shared treatment planning and target intervention strategies.

ELIGIBILITY:
Patient Inclusion Criteria:

1. Adult (> 18 years) English speaking patients
2. Treated with curative intent with chemo-radiotherapy
3. Seen in routine clinic follow-up within 5 years post completion of treatment

Patient Exclusion Criteria:

1. Patients at their anticipated last clinic visit prior to cancer center discharge
2. Patients unable to complete the EORTC QLQ CX-24 questionnaire due to inability to read or write.
3. Non-English speaking patients
4. Patients of the principal investigator. The rationale for this is that patients of the principal investigator who complete the Feedback form may be biased and this may be reflected in the results.

Oncologist Inclusion Criteria:

1. Oncologists who treat cervix cancer
2. Oncologists with at least one consenting patient enrolled in the study

Oncologist Exclusion Criteria:

1) Principal investigator listed on the protocol. The rationale for this is that oncologists who are also investigators on this study may have inherent bias in the study which may be reflected in the results of the Feedback form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cervical cancer patients seen in follow-up, up to 5-years post-treatment, at the Princess Margaret, Odette, and Royal Victoria Regional Health Center as well their treating Oncologists.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2020-05-25 (Actual); Study Completion 2020-05-25 (Actual)

PRIMARY OUTCOMES:
Percentage of EORTC QLQ CX24 questionnaire completed | 9 months
  Gather information on feasibility of administering questionnaire
Percentage of favorable scores (Agree or strongly agree) on Feedback Form | 9 months
  Gather information on acceptability of incorporating the questionnaire in routine follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Croke, MD, Principal Investigator — The Princess Margaret Cancer Foundation
Locations (3):
- Canada (3):
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario